CLINICAL TRIAL: NCT03890965
Title: Effects of the Application of a Reflex Locomotion Program on Sitting in the Neurological Hand of the Chronic Adult Patient
Brief Title: Effects of the Application of a Reflex Locomotion Program in the Neurological Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NUMEN Foundation (Other)
Responsible Party: Principal Investigator, Luis Perales Lopez, Physiotherapy service coordinator, NUMEN Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NUMEN1
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Neurological Disorder
Keywords: stroke; Physical therapy; neurological hand; Vojta therapy
MeSH Terms: conditions — Nervous System Diseases; Stroke

STUDY DESIGN:
Intervention Model Description: Pretest-posttest trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Adult patients with chronic sequelae in the upper limb after neurological damage
  Interventions: Other: Reflex locomoction therapy

INTERVENTIONS:
Other: Reflex locomoction therapy — The intervention of the stimulation of the reflex locomotion is carried out in this study in a sitting position in a conventional chair, an unorthodox posture in the usual treatment of Vojta therapy.
  The reflex stimulation is performed by the passive pressure exerted by the weight of the wrist (pisiform) on the rubber sphere. Simultaneously the patient has to exert a slight pressure with the heel towards the ground with his foot. This foot will be the opposite of the wrist that has the sphere under the pisiform.
  Alternating each diagonal 4 times, 5 minutes each. Total session 20 minutes, 2 times x day, every day according to degree of affectation.

SUMMARY:
The recovery of the function of the hand is one of the most important aspects for patients who have suffered the consequences of neurological damage. Currently there are numerous therapeutic procedures aimed at rehabilitation that have scientific evidence such as restrictive therapy. However, dysfunction of the upper limb has an impact on the whole body that is not always taken into consideration.

DETAILED DESCRIPTION:
The intervention of the stimulation of the reflex locomotion is carried out in this study in a sitting position in a conventional chair, an unorthodox posture in the usual treatment of Vojta therapy.

Description of the sitting posture: the back in axial extension with the shoulders located in front of the hips.

The elbows must be supported with the medial epicondyl in contact on a table, whose height is at the level of the end of the patient's sternum.

The forearms are placed prone with the palms facing the surface. In this position we place a rubber sphere 3 centimeters in diameter under the pisiform of one of the patient's wrists.

The reflex stimulation is performed by the passive pressure exerted by the weight of the wrist (pisiform) on the rubber sphere. Simultaneously the patient has to exert a slight pressure with the heel towards the ground with his foot. This foot will be the opposite of the wrist that has the sphere under the pisiform.

It is a cross-stimulation, that is, pisiform in one hand together with the load in the heel of the opposite side.

Alternating each diagonal 4 times, 5 minutes each. Total session 20 minutes, 2 times per day, every day according to degree of affectation

The duration of the study will depend on the degree of involvement: mild 2 weeks, moderate 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Sequelae in the upper limb after neurological damage.
* Understanding and oral expression preserved.
* More than a year after the episode.
* Possibility of walking

Exclusion Criteria:

* Aphasia.
* Concomitant diseases: Diabetes and arthritis of the hand.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
kinesiological test of the upper limb | 2 weeks for mild grade and 3 months for moderate degree
  Shoulder: flexion and maximum abduction. Forearm: Supination / pronation. Wrist: maximum dorsal flexion. Hand: finger extension
The Box and Block Test | 2 weeks for mild grade and 3 months for moderate degree.
  The Box and Block Test is a functional outcome measure that is commonly used across multiple clinical populations due to its benefits of ease and speed of implementation; reliable, objective measurement; and repetition of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Perales Lopez, Doctor, Principal Investigator — NUMEN Foundation
Locations (1):
- NUMEN Foundation, Madrid, España, Spain